CLINICAL TRIAL: NCT04909021
Title: Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation Phase 1c Study to Evaluate the Safety and Immunogenicity of an Intranasal Live Attenuated Respiratory Syncytial Virus Vaccine (MV-012-968) in Seronegative Children 6-36 Months
Brief Title: Safety and Immunogenicity of an Intranasal Vaccine for Respiratory Syncytial Virus in Seronegative Children 6-36 Months
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meissa Vaccines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: MV-006
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: live attenuated vaccine; safety; immunogenicity; Phase 1 clinical trial; Pediatric; seronegative; children

STUDY DESIGN:
Intervention Model Description: 1st 5 subjects will be in Group 1 and randomized to investigational vaccine (IP) Dosage 1 or placebo. Safety Monitoring Committee (SMC) will review Group 1 data to Day 15 to allow dose escalation. Next 10 subjects will be in Group 2 and randomized to IP Dosage 2 or placebo. SMC will review Group 2 data to Day 15 to allow dose escalation. Next 12 enrolled subjects will be in Group 3 and randomized to IP Dosage 3 or placebo. SMC will review Group 3 data to Day 15 to allow dose escalation. Next 12 subjects will be in Group 4 and randomized to IP Dosage 4 or placebo. SMC will review Group 4 data to Day 15 to allow dose escalation. Next 12 subjects will be in Group 3a and randomized to IP Dosage 3 or placebo; if meet criteria will receive 2nd dose IP or placebo 28 days after 1st dose. Final 12 subjects will be in Group 4a and randomized to IP Dosage 4 or placebo; if meet criteria will receive 2nd dose IP or placebo 28 days after 1st dose.
Who Masked: Participant
Masking Description: The study is single-mask. Study participants and their parent(s)/guardian(s) will not know their child's study assignment; investigators, site staff, and site pharmacists will remain unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dosage Group 1: RSV Vaccine Dosage 1 (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 1
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 1)
- Dosage Group 2: RSV Vaccine Dosage 2 (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 2
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 2)
- Dosage Group 3: RSV Vaccine Dosage 3 (Single-dose) (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 3
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 3; single-dose)
- Dosage Group 3a: RSV Vaccine Dosage 3 (Two-dose) (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 3 followed by a second identical dose of the investigational RSV vaccine 28 days later
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 3; two-dose)
- Placebo (Single-dose) (Placebo Comparator): Participants in this arm will receive a single intranasal dose of placebo
  Interventions: Other: Placebo (single-dose)
- Placebo (Two-dose) (Placebo Comparator): Participants in this arm will receive a single intranasal dose of placebo followed by a second identical dose of placebo 28 days later
  Interventions: Other: Placebo (two-dose)

INTERVENTIONS:
Biological: Investigational RSV vaccine MV-012-968 (Dosage 1) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 1: RSV Vaccine Dosage 1
Biological: Investigational RSV vaccine MV-012-968 (Dosage 2) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 2: RSV Vaccine Dosage 2
Biological: Investigational RSV vaccine MV-012-968 (Dosage 3; single-dose) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 3: RSV Vaccine Dosage 3 (Single-dose)
Biological: Investigational RSV vaccine MV-012-968 (Dosage 3; two-dose) — Single dose administered intranasally on Day 1, followed by an identical dose administered intranasally at the Day 29 study visit
  Arms: Dosage Group 3a: RSV Vaccine Dosage 3 (Two-dose)
Other: Placebo (single-dose) — Single dose administered intranasally on Day 1
  Arms: Placebo (Single-dose)
Other: Placebo (two-dose) — Single dose administered intranasally on Day 1, followed by an identical dose administered intranasally at the Day 29 study visit
  Arms: Placebo (Two-dose)

SUMMARY:
This study evaluates an investigational vaccine that is designed to protect humans against infection with respiratory syncytial virus (RSV) and is administered as a nasal spray. Specifically, the study analyzes the safety of, and the immune response to, the vaccine when administered to healthy children between the ages of 6 and 24 months who are seronegative to RSV.

ELIGIBILITY:
Key Inclusion Criteria:

1. Children aged 6-36 months
2. Good health based on history, physical examination, and medical record review, without evidence or suspicion of chronic disease
3. Seronegative to RSV, as defined by serum nAb titer below the threshold described in the study protocol and operations manual
4. Written informed consent provided by parent(s)/guardian(s)

Key Exclusion Criteria:

1. Known or suspected chronic illness, particularly cardiopulmonary (including asthma or reactive airways disease), genetic or metabolic, hepatic, renal, infectious (including recurrent or chronic sinusitis), or immunodeficiency
2. Prior lab-confirmed RSV infection
3. Household or close contact (including but not limited to daycare) during the 21 days post-inoculation with anyone < 6 months old or immunocompromised (applies to first study inoculation)
4. Nasal obstruction (including due to anatomic/structural causes, acute or chronic rhinosinusitis, or other causes)
5. Receipt of immunoglobulins, monoclonal antibodies and/or any blood products, or ribavirin within 6 months prior to study inoculation, or planned use during study period
6. Receipt of an investigational RSV vaccine at any time
7. Any other condition that, in the judgment of the investigator, would be a risk to subject's safety and/or may interfere with study procedures or interpretation of results

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events (AEs) | Immediate post-vaccination period
  Frequency of solicited AEs will be measured, categorized by severity. Solicited AEs are predefined AEs that may occur after investigational vaccine administration
Unsolicited AEs | Immediate post-vaccination period
  Frequency of unsolicited AEs will be measured, categorized by severity. Unsolicited AEs are any untoward medical occurrences in a participant administered the investigational vaccine, regardless of causal relationship to the investigational vaccine. Unsolicited AEs can include unfavorable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with the use of the investigational vaccine.
Serious adverse events (SAEs) | Full study duration, an average of 1 year
  Frequency of SAEs will be measured, categorized by vaccine-relatedness . SAEs are AEs, whether considered causally related to the investigational vaccine or not, that threaten life or result in any of the following: death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or congenital anomaly/birth defect.
Medically attended adverse events (MAEs) | Full study duration, an average of 1 year
  Frequency of MAEs will be measured, categorized by vaccine-relatedness. MAEs are AEs, whether considered causally related to the investigational vaccine or not, with unscheduled medically attended visits, such as urgent care visits, acute primary care visits, emergency department visits, or other previously unplanned visits to a medical provider. Scheduled medical visits such as routine physicals, wellness checks, 'check-ups', and vaccinations, are not considered MAEs.
Change in RSV-specific serum neutralizing antibody (nAb) titers (GMT) | Baseline through Day 28, an average of six (6) weeks
  Change in serum RSV-specific neutralizing antibody (nAb) titers will be measured per participant.

SECONDARY OUTCOMES:
Change in serum binding (RSV F-specific) Immunoglobulin G (IgG) concentrations | Baseline through Day 28, an average of six (6) weeks
  Change in serum binding (RSV F-specific) IgG concentrations will be measured per participant
Change in nasal mucosal binding (RSV F-specific) Immunoglobulin A (IgA) concentrations | Baseline through Day 28, an average of six (6) weeks
  Change in nasal mucosal binding (RSV F-specific) IgA concentrations will be measured per participant
Potential vaccine virus shedding after a single intranasal dose of MV-012-968: frequency | Intranasal inoculation through Day 22, an average of three (3) weeks
  Frequency of any post-vaccination shedding of vaccine virus (as detected by plaque assay) after a single intranasal dose of MV-012-968 will be measured per dosage group and overall.
Potential vaccine virus shedding after a single intranasal dose of MV-012-968: magnitude | Intranasal inoculation through Day 22, an average of three (3) weeks
  If post-vaccination shedding of vaccine virus is detected by plaque assay after a single intranasal dose of MV-012-968, peak viral titer (measured in plaque forming units, PFU) will be measured per dosage group and overall
Potential vaccine virus shedding after a single intranasal dose of MV-012-968: duration | Intranasal inoculation through Day 22, an average of three (3) weeks
  If post-vaccination shedding of vaccine virus is detected by plaque assay after a single intranasal dose of MV-012-968, duration of shedding (in days) will be measured per dosage group and overall.

OTHER OUTCOMES:
RSV-confirmed medically attended acute respiratory infection during peak RSV season following study inoculation | Approximately five (5) months duration during peak RSV season, adjusted for local epidemiology
  Frequency of RSV-confirmed medically attended acute respiratory infection during peak RSV season following study inoculation will be measured, categorized by severity.
RSV-confirmed medically attended acute lower respiratory infection | Approximately five (5) months duration during peak RSV season, adjusted for local epidemiology
  Frequency of RSV-confirmed medically attended acute lower respiratory infection during peak RSV season following study inoculation will be measured, categorized by severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Lieberman, MD, Study Director — Meissa Vaccines, Inc.
Locations (12):
- United States (12):
  - MedPharmics, Phoenix, Arizona
  - Paradigm Clinical Research, La Mesa, California
  - The Emory Children's Center, Atlanta, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - MedPharmics, Metairie, Louisiana
  - Meridian Clinical Research, Hastings, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, Binghamton, New York
  - Aventiv Research, Columbus, Ohio
  - Coastal Pediatric Research, Summerville, South Carolina
  - PanAmerican Clinical Research, Brownsville, Texas
  - Benchmark Research, San Antonio, Texas

REFERENCES:
- [Background] Stobart CC, Rostad CA, Ke Z, Dillard RS, Hampton CM, Strauss JD, Yi H, Hotard AL, Meng J, Pickles RJ, Sakamoto K, Lee S, Currier MG, Moin SM, Graham BS, Boukhvalova MS, Gilbert BE, Blanco JC, Piedra PA, Wright ER, Moore ML. A live RSV vaccine with engineered thermostability is immunogenic in cotton rats despite high attenuation. Nat Commun. 2016 Dec 21;7:13916. doi: 10.1038/ncomms13916. PMID 28000669